CLINICAL TRIAL: NCT05847153
Title: The Mindful and Self-Compassionate Care Program Aim 2
Brief Title: MASC: Reducing Stress for Caregivers
Acronym: MASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christine S. Ritchie, MD, MPH, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023P001130; 1R01AG078204-01 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease and Related Dementias; Dementia Alzheimers
Keywords: ADRD; Caregiver stress; Dementia; Alzheimer; Self-compassion
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: MASC is an intervention that includes evidence based skills of: 1) mindfulness; 2) compassion toward others and self; 3) behavioral management skills. MASC has 6 sessions delivered in a group format over secure live video with Zoom. Each session includes psychoeducation on program skills, skill practice, strategies to incorporate the skill into the caregiver experience, and strategies for sustained practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention arm will be comprised of:
  1. Six Virtual Group Sessions. The sessions will teach mindfulness, self-compassion and behavioral management skills.
  2. At Home Practice. After each group session, participants will have the opportunity to integrate the practices learned into their everyday life.
  Interventions: Behavioral: MASC

INTERVENTIONS:
Behavioral: MASC — The intervention arm will be comprised of:
  1. Six Virtual Group Sessions. The sessions will teach mindfulness, self-compassion and behavioral management skills.
  2. At Home Practice. After each group session, participants will have the opportunity to integrate the practices learned into their everyday life.

SUMMARY:
Building on limitations of prior research, the investigators proposed to develop the Mindful and Self-Compassionate Care Program (MASC) to help caregivers of persons with Alzheimer Disease and Related Dementias (ADRD) manage stress associated with the general caregiver experience including stress stemming from managing challenging patient behaviors. MASC teaches: (1) mindfulness skills; (2) compassion and self-compassion skills; and (3) behavioral management skills. MASC also provides psychoeducation and group-based training and skill practice to facilitate skill uptake and integration within the caregiver experience and tasks.

DETAILED DESCRIPTION:
Over half of Alzheimer Disease and Related Dementias (ADRD) caregivers are actively looking for non-pharmacological interventions to decrease caregiver stress. Available programs do not meet the psychological and practical needs of stressed caregivers of persons with ADRD; better solutions are needed. First, while helpful, most support groups do not systematically teach behavioral management skills which caregivers report needing in order to manage challenging patient behaviors. Second, behavioral management skills interventions exist, but do not teach: 1) emotional regulation skills which are necessary in order to foster caregiver ability to access and use these skills to manage patient behaviors, and/or 2) self-compassion and compassion skills which are necessary to bypass guilt and loneliness and navigate behavioral symptoms which are common caregiver challenges. Third, mindfulness and self-compassion interventions are effective solutions for managing stress, and distress across multiple populations, but engagement and efficacy among diverse ADRD caregivers are limited.

The guiding hypothesis of this proposal is that combining evidence-based mindfulness and self-compassion skills with behavioral management skills within a multi-component program increases intervention potency and efficiently supports caregivers of persons with ADRD. Accounting for practical challenges to engagement (nr. sessions, delivery modality, skill practice) will also enhance uptake and reach.

The investigators will conduct an open pilot with exit interviews to explore feasibility benchmarks, target engagement and signal of improvement in stress, depression, anxiety and wellbeing (NIH stage 1A; N= up to 20 caregivers; N= up to 2 groups. Exit interviews will last 30 minutes and will be recorded, transcribed, and analyzed to refine study procedures. The investigators will use this information to revise and optimize MASC and our conceptual model, as needed to maximize feasibility and target engagement.

The investigators will recruit caregivers of persons with ADRD from local community organizations and caregiver support programs; dementia research programs; and from national programs that focus on caregiving.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English fluency and literacy
* Meeting criteria for being a caregiver (e.g., family or friend of a care recipient who provides unpaid care)
* Must live with and care for an individual with ADRD
* Must have been in a caregiver role for more than 6 months
* Must provide an average 4 hours of supervision or direct assistance per day for the are recipient
* Perceived Stress Scale-4 (4-item) version >=6
* Had managed 1 or more behavioral symptoms in past month

Exclusion Criteria:

* Recent change ini psychotropic treatment for depression or anxiety
* Use of mindfulness apps or any meditation (more than 60 min/week in past 6 months)
* Involvement in another clinical trial for caregivers, a score >= 4 on the Portable Mental Status Questionnaire (PMSQ)
* No stated concerns or distress related to care recipient's disruptive behaviors
* Involvement in another clinical trial for caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine S Ritchie, MD, MSPH, Principal Investigator — Massachusetts General Hospital; Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jutkowitz E, Kane RL, Gaugler JE, MacLehose RF, Dowd B, Kuntz KM. Societal and Family Lifetime Cost of Dementia: Implications for Policy. J Am Geriatr Soc. 2017 Oct;65(10):2169-2175. doi: 10.1111/jgs.15043. Epub 2017 Aug 17. PMID 28815557
- [Background] Roche V. The hidden patient: addressing the caregiver. Am J Med Sci. 2009 Mar;337(3):199-204. doi: 10.1097/MAJ.0b013e31818b114d. PMID 19282676
- [Background] Sorensen S, Conwell Y. Issues in dementia caregiving: effects on mental and physical health, intervention strategies, and research needs. Am J Geriatr Psychiatry. 2011 Jun;19(6):491-6. doi: 10.1097/JGP.0b013e31821c0e6e. No abstract available. PMID 21502853
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Jennings LA, Reuben DB, Evertson LC, Serrano KS, Ercoli L, Grill J, Chodosh J, Tan Z, Wenger NS. Unmet needs of caregivers of individuals referred to a dementia care program. J Am Geriatr Soc. 2015 Feb;63(2):282-9. doi: 10.1111/jgs.13251. PMID 25688604
- [Background] Alsubaie M, Abbott R, Dunn B, Dickens C, Keil TF, Henley W, Kuyken W. Mechanisms of action in mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR) in people with physical and/or psychological conditions: A systematic review. Clin Psychol Rev. 2017 Jul;55:74-91. doi: 10.1016/j.cpr.2017.04.008. Epub 2017 Apr 23. PMID 28501707
- [Background] Pedro J, Monteiro-Reis S, Carvalho-Maia C, Henrique R, Jeronimo C, Silva ER. Evidence of psychological and biological effects of structured Mindfulness-Based Interventions for cancer patients and survivors: A meta-review. Psychooncology. 2021 Nov;30(11):1836-1848. doi: 10.1002/pon.5771. Epub 2021 Jul 28. PMID 34288218
- [Background] Conversano C, Orru G, Pozza A, Miccoli M, Ciacchini R, Marchi L, Gemignani A. Is Mindfulness-Based Stress Reduction Effective for People with Hypertension? A Systematic Review and Meta-Analysis of 30 Years of Evidence. Int J Environ Res Public Health. 2021 Mar 11;18(6):2882. doi: 10.3390/ijerph18062882. PMID 33799828
- [Background] Al-Refae M, Al-Refae A, Munroe M, Sardella NA, Ferrari M. A Self-Compassion and Mindfulness-Based Cognitive Mobile Intervention (Serene) for Depression, Anxiety, and Stress: Promoting Adaptive Emotional Regulation and Wisdom. Front Psychol. 2021 Mar 22;12:648087. doi: 10.3389/fpsyg.2021.648087. eCollection 2021. PMID 33828514
- [Background] Mahaffey BL, Mackin DM, Vranceanu AM, Lofaro L, Bromet EJ, Luft BJ, Gonzalez A. The Stony Brook Health Enhancement Program: The development of an active control condition for mind-body interventions. J Health Psychol. 2020 Nov-Dec;25(13-14):2129-2140. doi: 10.1177/1359105318787024. Epub 2018 Jul 16. PMID 30010422
- [Background] Lancaster GA. Pilot and feasibility studies come of age! Pilot Feasibility Stud. 2015;1(1):1. doi: 10.1186/2055-5784-1-1. Epub 2015 Jan 12. PMID 29611687
- [Derived] Travis A, O'Donnell A, Giraldo-Santiago N, Stone SM, Torres D, Adler SR, Vranceanu AM, Ritchie CS. Intervention for the Management of Neuropsychiatric Symptoms to Reduce Caregiver Stress: Protocol for the Mindful and Self-Compassion Care Intervention for Caregivers of Persons Living With Dementia. JMIR Res Protoc. 2024 Oct 11;13:e58356. doi: 10.2196/58356. PMID 39392675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.38 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Perceived Stress Scale (PSS-10) [Mean (Standard Deviation); unit: units on a scale] | 21.62 (7.07)
Neuropsychiatric Inventory Questionnaire (NPIQ) [Mean (Standard Deviation); unit: units on a scale] — Each of the 12 NPI-Q domains contains a survey question that reflects cardinal symptoms of that domain. Initial responses to each domain question are "Yes" (present) or "No" (absent). If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale. Presence range 0-12, 0 being not symptomatic. Severity range 12-36, 12 being mild. Distress range 0-60, 0 is not distressing.
  units on a scale
    NPI- Presence | 7 (2.71)
    NPI- Severity | 13.92 (6.87)
    NPI-Distress | 17.54 (10.32)
Center For Epidemiologic Studies Depression Scale [Mean (Standard Deviation); unit: units on a scale] | 22.15 (13.08)
Interpersonal Support Evaluation List [Mean (Standard Deviation); unit: units on a scale] | 35.62 (7.1)
UCLA Loneliness Scale [Mean (Standard Deviation); unit: units on a scale] | 6.08 (1.89)
Positive Affect Index [Mean (Standard Deviation); unit: units on a scale] | 40.92 (10.17)
Self-Compassion Scale Short Form [Mean (Standard Deviation); unit: units on a scale] — This scale measures the level of self-compassion a participant has towards themselves with 12 questions on a scale of 1-5 (1 meaning "almost never" and 5 meaning "almost always). Scores are mainly used in a comparative manner to examine outcomes for people scoring higher or lower in self-compassion. As an ad hoc rubric, you can consider scores 1.0-2.49 to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high. When trying to determine whether self-compassion levels are high or low relevant to a particular sample, some researchers use a median split.
  units on a scale | 3.06 (0.70)
Applied Mindfulness Process Scale Amps [Mean (Standard Deviation); unit: units on a scale] | 34.54 (7.92)
Compassion Scale [Mean (Standard Deviation); unit: units on a scale] — The Compassion Scale measures how much compassion one has for others with 16 questions. The highest score possible is a 5, meaning higher compassion, and the lowest score possible is a 2, meaning lower compassion.
  units on a scale | 4.23 (0.52)
Revised Scale For Caregiving Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — This scale measures how confident participants are that they can keep up with their own activities and also respond to caregiving situations. There are 10 questions, rated 0 to 100, where 0 is not confident at all and 100 is very confident. The score is calculated by standardizing each score from 0-10 and summing the total. A 0 is the minimum, meaning not confident, and 100 is the maximum, meaning very confident.
  units on a scale | 56.85 (12.99)
WHO-5 Wellbeing Index [Mean (Standard Deviation); unit: units on a scale] — The Who-5 well-being scale measures perceived quality of life. The raw score is calculated by totaling the scores of the five questions. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
  units on a scale | 12.23 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment
Description: The investigators will examine feasibility of recruitment overall. The investigators will report proportion of eligible participants who are eligible and choose to enroll in the study. The investigators will also explore the percent of racial and ethnically diverse participants across the entire sample. Benchmark: ≥70% of participants who are eligible will enroll; ≥38% of participants are racial and ethnic minorities (US representation)
Time Frame: Baseline
Population: 16 participants were eligible and 13 chose to enroll. Out of the 13 that chose to enroll, 4 were racial and ethnic minorities.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 16
Participants
  Enrolled Participants | 13
  Racial and Ethnic Minorities: number analyzed (Participants) | 13
  Racial and Ethnic Minorities | 4

2. Primary Outcome: Number of Participants With Less Than 25% of Missing Questionnaires at Baseline
Description: The investigators will calculate the proportion of participants completing the study who have less than 25% of missing questionnaires. Benchmark: ≥70% participants will have less than 25% missing questionnaires.
Time Frame: Baseline
Population: The number of participants who completed the baseline questionnaire is 13.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 13
Participants | 13

3. Primary Outcome: Number of Participants With Less Than 25% of Missing Questionnaires at Post-Intervention
Description: as for outcome 2
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: While 13 participants completed the baseline survey, only 12/13 participants attended the sessions (intervention). Therefore,12 participants were counted as completing the study, which was measured as those who completed the baseline survey and attended the intervention sessions. 11/12 completed participants completed the post-intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 12
Participants | 11

4. Primary Outcome: Number of Participants With no Questionnaries Missing Fully at Baseline
Description: The investigators will assess the feasibility of the quantitative measures sent to participants. Benchmark: No questionnaires missing fully in ≥25% participants.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 13
Participants | 13

5. Primary Outcome: Number of Participants With no Questionnaries Missing Fully at Post-intervention
Description: as for outcome 4
Time Frame: Post-intervention (6-8 weeks post baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 13
Participants | 11

6. Other Pre Specified Outcome: Symptoms of Depression
Description: The investigators will use the Center for Epidemiological Studies-Depression Scale (CES-D). This is a 20-item scale widely used with ADRD participants. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time) In scoring the CES-D, possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 22.15 (13.08)

7. Other Pre Specified Outcome: Symptoms of Depression
Description: as for outcome 6
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 11/13 participants completed the post-intervention CES-D survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale | 16 (9.27)

8. Other Pre Specified Outcome: Mindfulness
Description: The investigators will use the Five Facets Mindfulness Questionnaire (FFMQ) to assess caregivers mindfulness based on 5 subscales (observing, describing, awareness, non-judging, non-reactivity). Average scores are calculated by summing the responses and dividing by the number of items, and indicate the average level of agreement with the each subscale (1 = rarely true, 5 = always true). Higher scores are indicative of someone who is more mindful in their everyday life. Its facet scores range from 3-15.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mindfulness
Description: as for outcome 8
Time Frame: Post-intervention (6-8 weeks post baseline)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Perceived Stress Scale
Description: The investigators will use the Perceived Stress Scale 10 (PSS-10) to assess perceived stress using a 5-point Likert scale.
  Scoring Instructions: Total score is determined by adding together the scores of each of the four items. Questions 2 and 3 are reverse coded. Questions 1 and 4: 0 = Never; 1 = Almost never; 2 = Sometimes; 3 = Fairly often; 4 = Very often Questions 2 and 3: 4 = Never; 3 = Almost never; 2 = Sometimes; 1 = Fairly often; 0 = Very often.
  Scores range from 0 to 40 with higher scores indicating more stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 21.62 (7.07)

11. Other Pre Specified Outcome: Perceived Stress Scale
Description: as for outcome 10
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 11/13 participants completed the post-intervention PSS-10 survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale | 16.91 (4.44)

12. Other Pre Specified Outcome: Symptoms of Anxiety
Description: The investigators will use State Trait Anxiety Inventory (STAI) state subscales (20 items) to assess anxiety symptoms in response to stressful situations. STA has been successfully used with ADRD participants.
  The range of possible scores varies from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Time Frame: Baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Symptoms of Anxiety
Description: as for outcome 12
Time Frame: Post-intervention (6-8 weeks post baseline)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: The Self-Compassion Scale
Description: The Self-Compassion Scale - Short Form (SCS-SF) is a 12-item self-report measure that is used by adults to measure their capacity for self-compassion - the ability to hold one's feelings of suffering with a sense of warmth, connection and concern. Self-Kindness Items: 2, 6 Self-Judgment Items (Reverse Scored): 11, 12 Common Humanity Items: 5, 10 Isolation Items: 4, 8 Mindfulness Items: 3, 7 Over-identification Items : 1, 9 = max score of 8 per category
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 3.06 (0.7)

15. Other Pre Specified Outcome: The Self-Compassion Scale
Description: as for outcome 14
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the post-intervention SCS survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 3.35 (0.70)

16. Other Pre Specified Outcome: Compassion
Description: The Compassion Scale (CS) has 16 items assessing common humanity, kindness toward others and ability to understand the suffering or challenges of others. Kindness items: 2, 6, 10, 14 Common Humanity items: 4, 8, 12, 16 Mindfulness items: 1, 5, 9, 13 Indifference items (reverse scored): 3, 7, 11, 15. Subscale scores are computed by calculating the mean of the four subscale item responses. To compute a total compassion score, reverse score the indifference items then take a grand mean of all items. When examining subscale scores, higher scores on indifference items indicate less compassion before reverse-coding, and more compassion after reverse coding. Participants can choose to report indifference scores with or without reverse-coding, but items must be reverse coded before calculating a total compassion score.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 4.23 (0.52)

17. Other Pre Specified Outcome: Compassion
Description: as for outcome 16
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the CS post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 4.16 (0.59)

18. Other Pre Specified Outcome: Caregiver Self-efficacy
Description: This scale measures how confident participants are that they can keep up with their own activities and also respond to caregiving situations. There are 10 questions, rated 0 to 100, where 0 is not confident at all and 100 is very confident. The score is calculated by standardizing each score from 0-10 and summing the total. A 0 is the minimum, meaning not confident, and 100 is the maximum, meaning very confident.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 56.85 (12.99)

19. Other Pre Specified Outcome: Caregiver Self-efficacy
Description: as for outcome 18
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 9/13 participants completed the RSCSE post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
score on a scale | 58.33 (15.72)

20. Other Pre Specified Outcome: Loneliness
Description: The University of California, Los Angeles (UCLA) 3-item loneliness scale assess relational connectedness, social connectedness and self-perceived isolation.
  The scores for each individual question can be added together to give participants a possible range of scores from 3 to 9. Researchers in the past have grouped people who score 3 - 5 as "not lonely" and people with the score 6 - 9 as "lonely".
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 6.08 (1.89)

21. Other Pre Specified Outcome: Loneliness
Description: as for outcome 20
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 11/13 participants completed the UCLA post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale | 5.91 (1.81)

22. Other Pre Specified Outcome: Social Support
Description: Interpersonal Support Evaluation List short form (ISEL) has 12 items assessing appraisal, belonging and tangible social support.
  A 12-item measure of perceptions of social support. Response options range from 1-4 with 4 = "definitely true" if the participant is sure it is true about them, 3= "probably true" if the participant thinks it is true but is not absolutely certain. Similarly, the participant should circle 1 = "definitely false" if they are sure the statement is false and 2 = "probably false" if the participant thinks it is false but is not absolutely certain. This questionnaire has three different subscales designed to measure three dimensions of perceived social support. These dimensions are: 1.) Appraisal Support 2.) Belonging Support 3.) Tangible Support Each dimension is measured by 4 items on a 4-point scale ranging from "Definitely True" to "Definitely False". The minimum score is 12 and the maximum is 48. Higher scores are a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 35.62 (7.10)

23. Other Pre Specified Outcome: Social Support
Description: A 12-item measure of perceptions of social support. Response options range from 1-4 with 4 = "definitely true" if the participant is sure it is true about them, 3= "probably true" if the participant thinks it is true but is not absolutely certain. Similarly, the participant should circle 1 = "definitely false" if they are sure the statement is false and 2 = "probably false" if the participant thinks it is false but is not absolutely certain. This questionnaire has three different subscales designed to measure three dimensions of perceived social support. These dimensions are: 1.) Appraisal Support 2.) Belonging Support 3.) Tangible Support Each dimension is measured by 4 items on a 4-point scale ranging from "Definitely True" to "Definitely False". The minimum score is 12 and the maximum is 48. Higher scores are a better outcome.
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 11/13 participants completed the ISEL post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale | 37.73 (6.37)

24. Other Pre Specified Outcome: Well-being
Description: World Health Organization-Five Well-Being Index (WHO-5) has 5 items assessing emotional well-being.
  The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life The outcome measure represents the mean of the raw score.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 12.23 (4.25)

25. Other Pre Specified Outcome: Well-being
Description: as for outcome 24
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 9/13 participants complete the WHO post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
score on a scale | 15 (4.27)

26. Other Pre Specified Outcome: Distress Due to Patient Challenges Behaviors
Description: The Neuropsychiatric Inventory Caregiver Distress Scale has 12 items assessing distress associated with dementia patient's behaviors such as apathy, elation, disinhibition. Participant distress is rated for each positive neuropsychiatric symptom domain on a scale anchored by score from 0 to 5 points. The Score is: 0 = Not distressing at all, 1 = Minimal (slightly distressing, not a problem to cope with), 2 = Mild (not very distressing, generally easy to cope with), 3 = Moderate (fairly distressing, not always easy to cope with), 4 = Severe (very distressing, difficult to cope with), 5 = Extreme of Very Severe (extremely distressing, unable to cope with). The minimum is 0, indicating less distress and a better outcome and he maximum is 60, indicating more distress and a worse outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 17.54 (10.32)

27. Other Pre Specified Outcome: Distress Due to Patient Challenges Behaviors
Description: as for outcome 26
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 11/13 participants completed the NPI distress post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale | 15.55 (7.92)

28. Other Pre Specified Outcome: Satisfaction With the Intervention
Description: The investigators will use the Client Satisfaction Questionnaire (CSQ-3) to assess participants' satisfaction with the intervention. The questionnaire consists of 3 questions rating participants' satisfaction on a scale of 1-4, with 1 being not satisfied at all and 4 being very satisfied. Total possible score is 12 and the least possible score is 3.
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the CSQ post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 10.5 (1.9)

29. Other Pre Specified Outcome: Patient's Global Impression of Change (PGIC)
Description: The investigators will ask participants about their perceptions of whether or not they feel that they improved in stress, depression, anxiety and wellbeing. PGIC is a 5 point scale depicting a participant's rating of overall improvement. Participants rate their change as "much improved", "minimally improved", "no change", "minimally worse", or "much worse". A score of 1 is much worse and 5 is much improved.
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the PGIC post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 4.4 (0.70)

30. Other Pre Specified Outcome: Therapist Fidelity
Description: The investigators will assess both therapists' ability to deliver the content of each session (through therapist completed adherence checklists) and therapist fidelity (through independent review of recorded sessions by Co-Investigator). Ratings will be given for each of six sessions on the following scale: 1=Not Present,3=Slightly Present,5=Moderately Present,7=Often Present,10=Always Present. An average score of 10 for all sessions represents all content always delivered, and an average score of 1 represents no content delivered as intended. Benchmark: >=75% of MASC sessions components delivered as intended; 20% sessions rated.
Time Frame: Baseline through Post-intervention (6-8 weeks post baseline)
Population: Both groups were analyzed with 6 sessions in each group. Number of participants in both sessions varied from 9-12.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Sessions
Arm/Group | Intervention
Number analyzed (Participants) | 12
Number analyzed (Sessions) | 60
score on a scale | 8.9 (0.47)

31. Other Pre Specified Outcome: Perceptions of Questionnaire Battery
Description: The investigators will use the 'Perceptions of Questionnaire Battery' qualitative measure to assess how appropriately the participants fill the questionnaires, address their perception of stress, emotional distress and all other questionnaires.
Time Frame: Post-intervention (6-8 weeks post baseline)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Adherence to Home Practice
Description: The investigators will report proportion of participants who complete weekly home practice.
Time Frame: Weekly (up to 5 weeks)
Population: 12/13 participants attended sessions and were sent homepractice surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 12
Participants
  Week 1 | 10
  Week 2 | 8
  Week 3 | 8
  Week 4 | 6
  Week 5 | 7

33. Other Pre Specified Outcome: Perceptions of Email and Text Reminders
Description: The investigators will assess participants' perception of emails and text messages reminders by asking, "Do participants think that the amount of emails/texts received was: too little, just enough, too much?"
Time Frame: Post-intervention (6-8 weeks post baseline)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Credibility and Expectancy
Description: The investigators will use the Credibility and Expectancy Questionnaire (CEQ) to assess participants' perceptions that the treatment will work after participating in the intervention. The CEQ utilizes two scales during the administration (1-9, and 0-100%), and so a composite score was derived for each factor (expectancy and credibility) by first standardizing the individual items and then summing those items for each factor. The minimum score is a 1, indicating worse outcome and less credibility and the maximum score is a 9, indicating a better outcome and more credibility.
Time Frame: Post-Intervention
Population: 9/13 participants filled out the post-intervention CEQ survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
score on a scale | 8 (0.71)

35. Other Pre Specified Outcome: Applied Mindfulness Process Scale
Description: The Applied Mindfulness Process Scale (AMPS) is a process measure used to quantify how participants in mindfulness-based interventions (MBIs) use mindfulness practice when facing challenges in daily life. Development and validation of the AMPS yielded 15 items representing three domains of applied mindfulness processes: (a) decentering, (b) positive emotional regulation, and (c) negative emotional regulation. Increases over time in AMPS scores suggest greater application of the use of mindfulness skills in daily life coinciding with mindfulness practice. Instructions for scoring:(1) Sum each factor individually to obtain a score ranging from 0-20, and/or (2) sum all 15 items to obtain a score ranging from 0-60. This is used as a replacement for the FFMQ.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 34.54 (7.92)

36. Other Pre Specified Outcome: Applied Mindfulness Process Scale
Description: as for outcome 35
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the post-intervention AMPS survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 38 (10.44)

37. Other Pre Specified Outcome: Modified Perception of Global Improvement
Description: The Modified Perception of Global Improvement (MPGI) is a global index designed to measure a participant's interpretation of changes in perceptions of stress following intervention. 0 indicates not improved and 1 indicates improved.
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 9/13 participants completed the MPGI post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
score on a scale | 0.89 (0.33)

38. Other Pre Specified Outcome: Positive Affect Index
Description: The Positive Affect Index (PAI) (5 items) assesses communication quality, closeness, similarity of views on life, engagement in joint activities and overall relationship quality. Each item is rated on a six-point scale and responses are summed for a total score. Possible scores range from 10 to 60 with higher scores indicating better relationship quality.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 40.92 (10.17)

39. Other Pre Specified Outcome: Positive Affect Index
Description: as for outcome 38
Time Frame: Post-intervention (6-8 weeks post baseline)
Population: 10/13 participants completed the PAI post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 38 (8.90)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant by participant self-report over the course of baseline administration (upto 1 week before the intervention started), the six week intervention, and up to the post-intervention assessment, which was conducted up to 1-week after conclusion of the intervention.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05847153/Prot_SAP_000.pdf